CLINICAL TRIAL: NCT03378414
Title: A Clinical Research on the Safety/Efficacy of Umbilical Cord Mesenchymal Stem Cells Therapy for Patients With Spinocerebellar Ataxia
Brief Title: Umbilical Cord Mesenchymal Stem Cells Therapy (19#iSCLife®-SA) for Patients With Spinocerebellar Ataxia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sclnow Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCLnow-XY-03
Record Dates: First submitted 2017-12-12; First posted 2017-12-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Spinocerebellar Ataxia Type 1; Spinocerebellar Ataxia Type 2; Spinocerebellar Ataxia Type 3; Spinocerebellar Ataxia Type 6
Keywords: Spinocerebellar Ataxia,Mesenchymal Stem Cells
MeSH Terms: conditions — Spinocerebellar Ataxias; Machado-Joseph Disease | interventions — Infusions, Intravenous; Injections, Spinal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intravenous infusion group (Experimental): Umbilical cord mesenchymal stem cells (SCLnow 19#)
  Interventions: Procedure: Intravenous infusion; Biological: umbilical cord mesenchymal stem cell
- Intrathecal injection group (Experimental): Umbilical cord mesenchymal stem cells (SCLnow 19#)
  Interventions: Procedure: Intrathecal injection; Biological: umbilical cord mesenchymal stem cell
- Control groups (No Intervention): No intervention

INTERVENTIONS:
Procedure: Intravenous infusion — Intravenous infusion of mesenchymal stem cells: 2 * 10^7 cells (30ml)
  Arms: Intravenous infusion group
Procedure: Intrathecal injection — Intrathecal injection of mesenchymal stem cells: 2 * 10^7 cells (1ml)
  Arms: Intrathecal injection group
Biological: umbilical cord mesenchymal stem cell — Treat patients with umbilical cord mesenchymal stem cell (SCLnow 19#), the dosage based on different procedure
  Arms: Intrathecal injection group; Intravenous infusion group

SUMMARY:
The purpose of this study is verify the safety and efficacy of Human Umbilical Cord Mesenchymal Stem Cells (UC-MSC) therapy for patients with Spinocerebellar Ataxia, and in addition, explore the possible mechanisms of UC-MSC therapy in Spinocerebellar Ataxia.

DETAILED DESCRIPTION:
This is a random, open label, and parallel controled experiment. 45 patients are selected and sign consent forms, then divided into three groups. Doctors collect the basic information of patient (including age,height, mental condition, vital sign, history of disease, pharmaco-history, genotype test, and so on.) All patients receive laboratory and image examination as baseline. Then, they will give cell treatment based on the clinical protocol. Doctors have follow-up visit on 1, 2, 3, 6, and 12 months after treatment, and do efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and genomic test diagnoses as spinocerebellar ataxias (SCA) (include SCA 1, SCA 2, SCA 3, SCA 6), SARA (Scale for Assessment and Rating of Ataxia) score is 2-5, can complete 8-meter walking test（8MW）
* Do not receive stem cells treatment in 6 months
* Participants sign the consent form based on the experiment process and statement

Exclusion Criteria:

* Cardiac, renal, hepatic insufficiency; total bilirubin is 1.5 times higher than normal value, aspartate transaminase（AST）or alanine aminotransferase（ALT）is 2.5 times higher than normal value
* Hemogram: total white blood cells <3.0 * 10^9 cells/L, blood platelet <75 * 10^9/L, hemoglobin <100g/L
* pneumonia, or severe infection
* With severe allergic history
* Brain organic disorder, like brain tumor
* Serum with HIV, syphilis antibody positive
* Severe mental disease, cognitive disorder patients
* Other severe system or organ organic disease
* Pregnant, breast feeding, or planning pregnant women
* Participate other clinical experiments in 3 months
* With some other conditions that doctor propose not to participate

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Scale for the assessment anf rating of ataxia (SARA) | 12 months
  Based on SARA score to calculate treatment efficacy. The equation is as follow, Efficacy = (patients who accepted treatment are effective/patients who accepted treatment)* 100% Effective: after 12 months, score of patient decrease 1 point or more; Ineffective: after 12 months, score decrease less than 1 point or increase.

SECONDARY OUTCOMES:
Image examinations | 12 months
  MRI plain scan of brain.
Inventory of Non-Ataxia Symptoms (INAS) score | 12 months
  Using Inventory of Non-Ataxia Symptoms (INAS) score to determine the presence and severity of non-ataxia signs.
Cerebrospinal fluid (csf) routine | 12 months
  Patients is observed by professionals, compare the changes of each observation point and baseline. Baseline is the data acquire from patients before stem cells treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jiang, Principal Investigator — Xiangya Hospital of Central South University